CLINICAL TRIAL: NCT01693211
Title: Prospective Evaluation of Circularity and Diameter of Femtosecond Laser Versus Manual Anterior Capsulotomy in Singapore National Eye Centre
Acronym: 1118
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1118
Record Dates: First submitted 2012-09-14; First posted 2012-09-26 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Primary Disease: Cataract
Keywords: femtosecond laser; cataract; control study; prospective
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Capsulorhexis and pre-fragmentation of the nucleus are performed by the femtosecond laser.
  Interventions: Device: Femtosecond Laser (VICTUS™ Femtosecond Laser Platform)
- Group B (Active Comparator): The Capulorhexis and nuclear fragmentation are performed manually.
  Interventions: Device: Manual (CCC technique with Utrata forceps)

INTERVENTIONS:
Device: Femtosecond Laser (VICTUS™ Femtosecond Laser Platform) — Capsulotomy and pre-fragmentation of the nucleus are performed by the femtosecond laser.
  Arms: Group A
Device: Manual (CCC technique with Utrata forceps) — Capsulorhexis and pre-fragmentation are performed manually.
  Arms: Group B

SUMMARY:
This is a prospective, randomized study evaluating the circularity of the anterior capsulotomy performed by the VICTUS femtosecond work station (Group A) versus the manual capsulotomy (Group B) of a minimum of 22 eyes and maximum of 30 eyes per group diagnosed with cataract, scheduled to undergo removal by phacoemulsification with intraocular lens implantation in SNEC.

The primary study end point is to determine if the circularity of the created rhexis is better in Group A as compared to Group B.

The secondary study end point is to determine the diameter of rhexis is more precise and reproducible in Group A as compared to Group B.

DETAILED DESCRIPTION:
This clinical study is a controlled, open, randomized, prospective, single-centre, single-surgeon eye study to determine the precision of intraocular cuts for anterior capsulotomy in connection to cataract surgery and IOL implantation. The cuts are applied by means of the VICTUS femtosecond laser system using a cylindrical cut pattern with diameter and height dependent on anterior chamber depth, pupil diameter and ocular lens size for Group A and the manual surgery technique for Group B.

The allocation of the surgery technique will be randomized between the study patient. Each surgery technique represents a study group. In Group A the anterior capsulotomy and lens fragmentation will be performed by means of femtosecond laser surgery. Group B acts as a control group where the capsulotomy as well as the lens fragmentation is performed manually.

The hypothesis of the study is that by means of intraocular, laser-induced cuts, circularity of the capsulotomy can be improved in a safe and effective way.

A detailed pre-operative examination will ensure that every interested and willing patient fulfils the inclusion criteria of this study. Post-operative examinations, which should document the success of the treatment, are to be carried out after 1-day, 1-week, 1-month.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients undergoing phacoemulsification and IOL implant surgery for cataract, the diagnosis of which has been confirmed by another investigator.
* Clear cornea media
* Pupil must be able to dilate to at least 6mm in diameter measured with the pupil gauge

Exclusion Criteria:

* Pre-existing posterior capsule rupture Difference between maximum and minimum K-values must not be more than 5 D. The maximum K- value may not exceed 60 D and the minimal value may not be smaller than 37 D.
* Corneal disease or pathology that precludes transmission of laser wavelength or distortion of laser light.
* Subjects with a poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally.
* Lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye.
* Patients with disorders of the ocular muscle, such as nystagmus or strabismus Keratoconus
* ACD < 1.8 mm or ACD > 4.5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Circularity of created rhexis | intraoperative
  The primary study end point is to determine if the circularity of the created rhexis is better in Group A as compared to Group B. On the day of surgery immediately after the creation of the rhexis via an recorded surgical video.

SECONDARY OUTCOMES:
Diameter of the created rhexis | intraoperative
  The secondary study end point is to determine the diameter of rhexis is more precise and reproducible in Group A as compared to Group B. On the day of surgery immediately after the creation of the rhexis via an recorded surgical video.

OTHER OUTCOMES:
Centration of the created rhexis relative to the pupil | surgery day, 1-Day, 1-week, 1-Month
  The additional outcome is to determine if the centration of the created rhexis relative to the pupil is better in Group A as compared to Group B. On the day of surgery immediately after the creation of the rhexis via an recorded surgical video and postoperative (1-Day, 1-week, 1-Month) based on slit lamp pictures.

CONTACTS AND LOCATIONS:
Overall Officials: Soon Phaik Chee, Assoc Prof, Principal Investigator — Singapore National Eye Center
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore, Singapore

REFERENCES:
- See also: Sponsor — http://www.technolaspv.com/